CLINICAL TRIAL: NCT01917682
Title: A Post-Market Registry for the Evaluation of the CorPath 200 System Effectiveness in Percutaneous Coronary Interventions
Brief Title: Post-Market CorPath Registry on the CorPath 200 System in Percutaneous Coronary Interventions
Acronym: PRECISION
Status: Completed | Type: Observational
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRECISION CorPath Registry
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: robotic-assisted PCI; coronary intervention; CorPath PRECISION Registry; PCI; angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Cohort: Subjects treated with CorPath-assisted Percutaneous Coronary Intervention (PCI)
  Interventions: Procedure: CorPath-assisted Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: CorPath-assisted Percutaneous Coronary Intervention — Robotic-assisted Percutaneous Coronary Intervention
  Other Names: Robotic-assisted Percutaneous Coronary Intervention

SUMMARY:
To collect data on the routine patterns of use, safety and effectiveness, including the clinical and technical performance of the CorPath 200 System, in the delivery and manipulation of coronary guidewires and stent/balloon catheters during PCI procedures.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, multi-center patient registry of the CorPath 200 System to examine its performance during PCI procedure and patient outcomes through 72 hours post-procedure or hospital discharge, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Patients with coronary artery disease undergoing Percutaneous Coronary Intervention (PCI) with the CorPath 200 system.
3. The subject or the legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Concurrent enrollment in another device or drug study protocol that specifically excludes concurrent enrollment or that prevents collection of data required in this registry (concurrent participation in another registry is not an automatic exclusion criterion for this study).
2. Failure/inability/unwillingness to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease and with the clinical indication for Percutaneous Coronary Intervention (PCI).
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giora Weisz, MD, Principal Investigator — Columbia University Medical Center/New York-Presbyterian Hospital; Chris Cain, Study Director — VP, Clinical Affairs
Locations (16):
- United States (15):
  - UC San Diego Medical Center, San Diego, California
  - Valley View Hospital, Glenwood Springs, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Orlando Regional Medical Center, Orlando, Florida
  - North Georgia Heart Foundation, Gainesville, Georgia
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Spectrum Health System, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center/New York-Presbyterian Hospital, New York, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Carolinas Medical Center - Northeast, Concord, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Sanford Health, Sioux Falls, South Dakota
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth Univ. Medical Center, Richmond, Virginia
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients that had a robotic-assisted PCI procedure.
Period: Overall Study
Arm/Group | Study Cohort
Started | 754
Completed | 754
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Cohort
Number analyzed (Participants) | 754
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 554

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success
Description: Less than 30% residual stenosis post PCI in the lesion(s) treated with the CorPath system, without in-hospital major adverse coronary events (MACE).
Time Frame: In-hospital (72-hours or discharge, whichever occurs first)
Population: Number of participants with complete data to assess clinical success.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 743
Participants | 723

2. Secondary Outcome: Number of Participants With In-hospital Major Adverse Coronary Events (MACE)
Description: The composite of death, myocardial infarction, and target vessel revascularization that occurs within 72 hours of the procedure or prior to hospital discharge, whichever occurs first, in a subject treated with the CorPath 200 System.
Time Frame: In-hospital (72-hours or discharge, whichever occurs first)
Population: Number of participants with complete data to assess In-hospital Major Adverse Coronary Events (MACE).
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 754
Participants | 6

3. Secondary Outcome: Number of Participants With an Adverse Event
Description: All Serious Adverse Events (SAEs) and Unanticipated Adverse Device Effects (UADEs) from the start of the CorPath procedure until the end of the study will be summarized.
Time Frame: In-hospital (72-hours or discharge, whichever occurs first)
Population: Number of participants with complete data to assess Adverse Events.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 754
Participants | 18

4. Other Pre Specified Outcome: Overall Procedure Time
Description: Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
Time Frame: During procedure
Population: Number of participants that had completed data to assess Overall procedure time.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Study Cohort
Number analyzed (Participants) | 722
min | 61.9 (28.3)

5. Other Pre Specified Outcome: PCI Procedure Time
Description: Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
Time Frame: During procedure
Population: Number of participants that had complete data to assess PCI procedure time.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Study Cohort
Number analyzed (Participants) | 696
min | 43.6 (23.1)

6. Other Pre Specified Outcome: Fluoroscopy and/or X-Ray Time
Description: As recorded by an X-Ray System utilized during the procedure.
Time Frame: During procedure
Population: Number of participants with complete data to assess fluoroscopy and/or X-Ray time.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Study Cohort
Number analyzed (Participants) | 753
min | 15.0 (8.4)

7. Other Pre Specified Outcome: Contrast Fluid Volume
Description: The amount of contrast fluid used (mL) during the procedure.
Time Frame: During procedure
Population: Number of partcipants with completed data to assess contrast fluid volume.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Study Cohort
Number analyzed (Participants) | 750
mL | 181.1 (90.8)

8. Other Pre Specified Outcome: Patient Radiation Exposure - Dose-Area-Product
Description: DAP (dose-area-product) as recorded during the procedure.
Time Frame: During procedure
Population: Number of participants that had completed data to assess patient radiation exposure. The overall number of participants analyzed in the DAP and Cumulative groups differ because of incomplete data recorded from the sites.
Measure: Mean (Standard Deviation); unit: mGy*cm2
Arm/Group | Study Cohort
Number analyzed (Participants) | 635
mGy*cm2 | 120861.3 (256522.9)

9. Other Pre Specified Outcome: Patient Radiation Exposure - Cumulative Dose
Description: Cumulative dose (mGy) as recored during the procedure.
Time Frame: During procedure
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | Study Cohort
Number analyzed (Participants) | 679
mGy | 1631.5 (3664.5)

10. Other Pre Specified Outcome: Number of Participants Who Had a Conversions to Manual Technique.
Description: The overall number of conversions from the robotic PCI to manual PCI will be captured to analyze the technical success of the device.
Time Frame: During procedure
Population: Number of conversions from the robotic PCI to manual PCI in participants with complete data.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 948
Participants | 99

11. Other Pre Specified Outcome: Visual Measurement of Lesion Length
Description: Visual estimate by clinical operator prior to delivery of PCI device(s).
Time Frame: During procedure
Population: Operator visual lesion length estimate.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Groups:
- Visual Estimate: Operator visual estimate of lesion length.
Arm/Group | Visual Estimate
Number analyzed (Participants) | 754
Number analyzed (Lesions) | 557
mm | 17.3 (9.8)

12. Other Pre Specified Outcome: CorPath Measurement of Lesion Length
Description: Robotic measurement of lesion length using the CorPath System performed by the Clinical Operator.
Time Frame: During procedure
Population: Lesion length measured with CorPath System.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: lesions
Arm/Group | Study Cohort
Number analyzed (Participants) | 754
Number analyzed (lesions) | 557
mm | 19.1 (10.6)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the index procedure though participant discharged from the hospital or 72-hours post procedure, whichever occurred first.
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/754
Serious Adverse Events (participants affected / at risk) | 18/754
Other Adverse Events (participants affected / at risk) | 0/754
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Cohort (N=754)
TRANSIENT BRADYCARDIA/HYPOTENSION (Cardiac disorders) | 1 (1)
FLUID RETENSION (Cardiac disorders) | 1 (1)
RECURRENT CHEST, RIGHT SHOULDER, RIGHT ARM PAIN (Cardiac disorders) | 1 (1)
ACUTE NAUSEA AND VOMITING (Gastrointestinal disorders) | 1 (1)
URINARY TRACT INFECTION (Renal and urinary disorders) | 1 (1)
DISSECTION DURING MANUAL PCI LESION #2 (Cardiac disorders) | 1 (1)
LEFT MAIN DISSECTION (Cardiac disorders) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ABRUPT VESSEL CLOSURE, DUE TO ANGIOPLASTY DISSECTION (Cardiac disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
PERI-PROCEDURAL MI; NSTEMI/NON QWAVE MI (Cardiac disorders) | 4 (4)
PEA ARREST (Cardiac disorders) | 1 (1)
ACUTE CEREBROVASCULAR ACCIDENT (CVA) (Nervous system disorders) | 1 (1)
CONTRAST DYE ALLERGIC REACTION; HYPOTENSION (Cardiac disorders) | 1 (1)
HEMATOCHEZIA (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No